CLINICAL TRIAL: NCT03441165
Title: Intraoperative Laxity Evaluation of Anterior Cruciate Ligament Reconstruction, Anterior Cruciate Ligament Revision and Meniscus Transplantation
Brief Title: Intraoperative Laxity Assessment of ACL Reconstruction, ACL Revision and MAT
Acronym: INTRA_KIN
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Prof, Istituto Ortopedico Rizzoli
Other Study IDs: INTRA_KIN
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Intraoperative Musculoskeletal Injury
Keywords: ACL; MAT; REVISION; LAXITY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: ligament reconstruction and meniscus transplantation — ACL reconstruction ACL revision MAT

SUMMARY:
Intraoperative knee laxity evaluation of patiente undergoing ACL reconstruction, ACL revision, MAT

DETAILED DESCRIPTION:
The study aims to include all thise patients who will undergo anterior cruciate ligament reconstruction, anterior cruciate ligament revision or meniscus transplantation. These patients will undergo an intraoperative kinematic evaluation (pre- and post-ligament reconstruction / meniscal transplantation). There is no follow-up because all the data necessary to carry out the study are obtained during the operating session. In particular, the pre- and post-intervention values (acquired intraoperatively) will be compared using both the surgical navigator and the KiRA system in order to evaluate the effect of the surgical procedure on the value of both static and dynamic laxity of the knee joint. Moreover, limited to the data acquired with the KiRA system, a comparison will be also made with the controlateral limb.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have provided written informed written consent
2. Patients aged 14 to 65
3. Patients undergoing reconstructive surgery of the anterior cruciate ligament or revision of anterior cruciate ligament surgery or meniscus transplantation. Patients unable to understand and want patients who have not signed informed consent

Exclusion Criteria:

1. Patients unable to understand and to want
2. Patients who have not signed informed consent

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to include all patients who will undergo anterior cruciate ligament reconstruction, anterior cruciate ligament revision or meniscus transplantation. These patients will undergo an intraoperative kinematic evaluation (pre- and post-ligament reconstruction / meniscal transplantation). There is no follow-up because all the data necessary to carry out the study are obtained during the operating session. In particular, the pre- and post-intervention acquired values (intraoperatively) will be compared both by the surgical navigator and by the KiRA system in order to evaluate the effect of surgery on the value of both static and dynamic laxity of the knee joint. Moreover, limited to the data acquired with the KiRA system, a comparison will also be made with the lateral limb.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Laxity Evaluation | intraoperative
  Laxity Evaluation will be performed using the intraoperative navigation system

SECONDARY OUTCOMES:
Dynamic Laxity Evaluation | intraoperative
  Laxity Evaluation will be performed using the KiRA device

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, Principal Investigator — stefano.zaffagnini@unibo.it
Locations (1):
- Stefano Zaffagnini, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided